CLINICAL TRIAL: NCT04311138
Title: The Effect of Community-based Reablement in Remote Areas
Brief Title: Effect of Community-based Reablement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CY Song (Other)
Responsible Party: Sponsor-Investigator, CY Song, assistant professor, National Taipei University of Nursing and Health Sciences
Organization: National Taipei University of Nursing and Health Sciences (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-060-B
Record Dates: First submitted 2020-03-12; First posted 2020-03-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Long Term Care
Keywords: reablement; community

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Experimental group receive a 10-wk diversified community-based reablement service.
  Interventions: Other: community-based reablement service
- Control group (Active Comparator): Control group receive a 10-wk multicomponent training.
  Interventions: Other: multicomponent training

INTERVENTIONS:
Other: community-based reablement service — Experimental group receive a 10-wk diversified community-based reablement service including group exercise, cognitive training, health education for 1.5 hours, and individualized reablement for 1.0 hour.
  Arms: Experimental group
Other: multicomponent training — control group receive a 10-wk multicomponent training including 1.5-hr group intervention (group exercise, cognitive training, and health education) and 1.0-hr placebo intervention.
  Arms: Control group

SUMMARY:
This study aims o investigate the effect of a diversified community-based reablement on motor function, cognitive function, performance in activities of daily living (ADL), and physical performance of older people living in remote areas. Older adults who are mobile but unstable were recruited from 6 public elderly day care centers in remote areas of the New Taipei City. Experimental group received a 10-wk diversified community-based reablement service including group exercise, cognitive training, health education for 1.5 hours, and individualized reablement for 1.0 hour, while control group received 1.5-hr group intervention and 1.0-hr placebo intervention. The de Morton Mobility Index (DEMMI), Saint Louis Mental Status Examination (SLUMS), Barthel Index (BI), Canadian Occupational Performance Measure (COPM), and the Short Physical Performance Battery (SPPB) including balance, gait speed, chair stand tests were evaluated twice before and after interventions. The results of the current study are expected to provide evidence in supporting a novel and diversified community-based reablement in remote areas.

ELIGIBILITY:
Inclusion Criteria:

* living in community and participating in public elderly day care centers in remote areas of the New Taipei City
* speaking with Chinese or Taiwanese
* DEMMI score of 39-67

Exclusion Criteria:

* diagnosed with moderate or severe cognitive impairment (CDR score of 2 or above)
* unable to understand or follow one step instruction

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2019-11-29 (Actual); Study Completion 2019-11-29 (Actual)

PRIMARY OUTCOMES:
Change in mobility function | baseline and 10 weeks
  de Morton Mobility Index (DEMMI)
Change in cognitive function | baseline and 10 weeks
  Saint Louis Mental Status Examination (SLUMS)
Change in performance in activities of daily living | baseline and 10 weeks
  Barthel Index (BI)
Change in occupational performance | baseline and 10 weeks
  Canadian Occupational Performance Measure (COPM)
Change in physical performance | baseline and 10 weeks
  Short Physical Performance Battery (SPPB)

CONTACTS AND LOCATIONS:
Overall Officials: ChenYi Song, Principal Investigator — National Taipei University of Nursing and Health Sciences
Locations (1):
- National Taipei University of Nursing and Health Sciences, Taipei, Taiwan